CLINICAL TRIAL: NCT05472636
Title: Clinical and Histopathological Evaluation of 41 Cases of Pediatric Granuloma Annulare
Brief Title: Evaluation of 41 Cases of Pediatric Granuloma Annulare
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Esra Koku Aksu, Assoc. Prof., Istanbul Training and Research Hospital
Other Study IDs: 97
Record Dates: First submitted 2022-07-15; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Granuloma Annulare
Keywords: Granuloma Annulare; Pediatric Dermatology; Pediatric Granuloma Annulare
MeSH Terms: conditions — Granuloma Annulare

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients under the age of 18 who were admitted to the dermatology outpatient clinic between 2008-2021 and diagnosed with granuloma annulare

SUMMARY:
INTRODUCTION: Granuloma annulare is a non-infectious, granulomatous disease that can affect children and adults. Although there are many studies examining adult patients, there are limited studies examining pediatric granuloma annulare cases. It is aimed to examine the demographic, clinical, and pathological features of pediatric granuloma annulare cases in this study.

MATERIALS and METHODS: This study was performed retrospectively in a single-center, tertiary dermatology hospital. Forty-one patients, under the age of 18 who were admitted to the dermatology outpatient clinic between 2008-2021 and diagnosed with granuloma annulare were scanned from the hospital database and patient photograph archive. Demographic characteristics, and clinical and histopathological features were evaluated.

DETAILED DESCRIPTION:
Granuloma annulare; is a non-infectious, granulomatous skin reaction with potential triggers that can affect the adult and pediatric age group. Diabetes mellitus, hyperlipidemia, and malignancy have been described in association with adult granuloma annulare cases. While there are studies on the clinical, pathological features and associated diseases in patients with adult granuloma annulare, a limited number of studies have been conducted on pediatric granuloma annulare patients. Therefore, clinical and histopathological evaluation of pediatric granuloma annulare cases was planned in our study.

This study was performed retrospectively in a single-center tertiary dermatology hospital. Patients under the age of 18 who were admitted to the dermatology outpatient clinic between 2008-2021 and diagnosed with granuloma annulare were scanned from the hospital database and patient photograph archive. Cases with uncertain diagnosis were not included in the study. Cases with dermatological findings recorded in detail and/or diagnosed histopathologically were included in the study. Demographic features, lesion localization, lesion characteristics (size, elementary lesion, color), involvement (localized/generalized), histopathological features, concomitant diseases, differential diagnoses in cases with histopathology, regression time and recommended treatments were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Being under 18 years old
* Having granuloma annulare
* Applying to the Istanbul Training and Research Hospital, Dermatology Outpatient Clinic between 2008-2021
* Consenting to participate in the study

Exclusion Criteria:

-Being over 18 years old

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients under the age of 18 who were admitted to the dermatology outpatient clinic between 2008-2021 and diagnosed with granuloma annulare
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the genders of the pediatric patients with granuloma annulare | day 0
  male, female
Evaluation of the ages of the pediatric patients with granuloma annulare | day 0
  age (year)
Evaluation of the concomitant diseases of the pediatric patients with granuloma annulare | day 0
  the concomitant diseases of the participants
Evaluation of the lesion localization of the pediatric patients with granuloma annulare | day 0
  head and neck, upper extremity, lower extremity, trunk
Evaluation of the lesion duration of the pediatric patients with granuloma annulare | day 0
  the time interval in between appearance of the lesion and diagnosis (month)
Evaluation of the lesion type of the pediatric patients with granuloma annulare | day 0
  papule, pustule, plaque, nodule
Evaluation of the mean size of the lesion | day 0
  diameter (cm)
Evaluation of the clinical involvement | day 0
  localized, generalized
Histopathological evaluation of the infiltration type of the pediatric patients with granuloma annulare | day 0
  neutrophilic, lymphocytic, lymphohistiocytic, eosinophil, mixed infiltrations
Histopathological evaluation of the infiltration pattern of the pediatric patients with granuloma annulare | day 0
  Interstitial, palisadic
Evaluation of epidermal findings | day 0
  regular/irregular, hyperkeratosis, acanthosis
Evaluation of depth of infiltrate | day 0
  superficial, medium, deep

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No